CLINICAL TRIAL: NCT00427986
Title: Diabetic Macular Oedema: Quantification of the Effect of Rising the Intracapillary Osmotic Pressure With Intravenous Galactose on the Retinal Thickness
Brief Title: Clinical Study of the Effect of Intravenous Galactose on Diabetic Macular Oedema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No sufficient increase in plasma osmolarity by galactose (one patient included)
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Dorte Nellemann, galactose
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetes; Macular oedema; Osmosis; Galactose; Intravenous; Retinal thickness; Starling
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Galactose

INTERVENTIONS:
Drug: Galactose, intravenous

SUMMARY:
The purpose of the present study is to examine, if retinal swelling in diabetic patients can be reduced by an intravenous injection of galactose.

DETAILED DESCRIPTION:
Macular oedema (swelling of the retina) is a leading cause of severe visual loss and blindness in patients with diabetes. The oedema is caused by fluid accumulation in the retinal tissue from leaking capillaries and leads to an increase in the retinal thickness. Optical Coherence Tomography (OCT) has become the primary technique to estimate the retinal thickness objectively, and the scans can be performed without any discomfort to the patient after dilation of the pupils.

According to the Starling equation, a general basic physiologic rule, specific factors influence the fluid transport between the capillaries and the surrounding tissue. One of these factors is the balance between the large molecules within the vessel lumen and the surrounding tissue, e.g. the osmotic pressure balance. By changing the osmotic balance some drugs can reduce the fluid content in the tissue by extracting water from the tissue to the vessel lumen. Such a drug is galactose.

In the present study we examine, if treatment with intravenous galactose can reduce the retinal thickness in diabetic macular oedema evaluated by OCT during a three-hour monitoring. Galactose (0.5 mg/mL) is administered as 1 mL galactose per kg body weight + 10% with a maximum of 80 mL, and injection time is 5 min. If reduction of the thickness with galactose is found, it then confirms the application of the Starling osmotic forces on diabetic macular oedema. In the same time span series of venous blood samples are taken for analysis of plasma osmolarity and electrolytes. The systemic blood pressure is also monitored as well as the capillary glucose level.

As diurnal variations in the retinal thickness estimates potentially can influence the results, the OCT measurements and blood samples are repeated on a second day for each participant, without treatment with galactose for comparison. The order of two visits is given by randomisation.

Interim analysis will take place after inclusion of 15 to 20 patients to evaluate the need for inclusion of 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* clinically significant macular oedema
* visual acuity of minimum 40 letters by the ETDRS procedure
* retinal thickness of at least 250 microns in the foveal region on three retinal maps of the fast protocol of the StratusOCT at baseline or at least 300 microns outside the foveal region
* 1 disc area of oedema within 3000 microns from the foveal center on three retinal maps of the fast protocol of the StratusOCT at baseline
* maximal blood pressure 160/90 mmHg (mean of three measurements)
* informed consent

Exclusion Criteria:

* other ocular diseases or treatments, that can cause or influence the macular oedema, including prior laser photocoagulation. Traction oedema is allowed.
* glaucoma
* media opacities that significantly impairs the light reflection while scanning
* Pregnancy
* severe heart, lung and/or renal insufficiency (judged by the primary investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Retinal thickness estimated by the fast protocol of the StratusOCT (0, 2, 4, 8, 10, 15, 20, 30, 60, 90, 120 and 180 min). | three hours

SECONDARY OUTCOMES:
Side effects during the three-hour examination period, to evaluate if caused by galactose per se or by an increase in intracapillary osmotic pressure. | Three hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Nellemann Thornit, MD, Principal Investigator — Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Nordre Ringvej 57, DK-2600 Glostrup, Denmark
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Nordre Ringvej 57,, Glostrup Municipality, Denmark